CLINICAL TRIAL: NCT01075672
Title: Outcomes of Cognitive Behavioral Therapy (CBT) Interventions Provided by Unlicensed Professionals in a General Hospital Setting
Brief Title: Outcomes of Cognitive Behavioral Therapy (CBT) Interventions Provided by Unlicensed Professionals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, PhD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009P002479
Record Dates: First submitted 2010-02-22; First posted 2010-02-25 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obsessive Compulsive Disorder; Body Dysmorphic Disorder; Tourette Syndrome; Trichotillomania; Panic Disorder; Social Phobia; Generalized Anxiety Disorder; Depression; Post-Traumatic Stress Disorder; Attention Deficit Hyperactivity Disorder; Eating Disorder; Specific Phobia; General Medical Condition
Keywords: OCD; BDD; Tourette syndrome; trichotillomania; Compulsive Skin Picking; panic disorder; social phobia; generalized anxiety disorder; depression; PTSD; ADHD; eating disorder; Specific Phobia
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Body Dysmorphic Disorders; Tourette Syndrome; Trichotillomania; Panic Disorder; Phobia, Social; Generalized Anxiety Disorder; Depression; Stress Disorders, Post-Traumatic; Attention Deficit Disorder with Hyperactivity; Feeding and Eating Disorders; Phobia, Specific; Excoriation Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- Behavioral Medicine with Cognitive Behavioral Therapy (Experimental): Participants enrolled in this arm of this study will be treated by the behavioral medicine interns with cognitive behavioral therapy focused on both their general health concerns and mental health concerns.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — The participant will then undergo a structured clinical interview with a supervised psychology intern/fellow, which will take approximately 1-3 hours over the course of 1-3 sessions. The initial assessment will be followed by up to 24 sessions of cognitive behavioral therapy tailored to their particular diagnosis (most diagnoses/problems require approximately 12 sessions, some require fewer, others require more). The length of treatment will depend on the primary diagnosis/ problem and the complexity and severity of the case. The clinician and patient will agree on a treatment plan after the initial evaluation, targeting a particular mental health or health related behavioral problem with Cognitive Behavioral Therapy. This treatment plan will include an agreed upon number of treatment sessions (up to 24).
  Other Names: CBT

SUMMARY:
To examine the effectiveness and clinical care outcomes of cognitive-behavioral therapy interventions at Massachusetts General Hospital (MGH).

DETAILED DESCRIPTION:
Cognitive behavioral interventions are the most widely studied and evidenced-based psychosocial treatment approaches for mental health and health related behavioral problems. Despite their documented efficacy, there is a scarcity of licensed mental health professionals who are available to treat patients with problems that would be amenable to Cognitive Behavioral Therapy (CBT). While CBT interventions have a strong base in terms of efficacy in randomized trials, effectiveness and dissemination studies are lacking in comparison, and hence, these interventions are not reaching the patients in most need of services. Complicating the problem further, insurance companies typically do not reimburse for services provided by trainees who are not licensed. This is a public mental health problem because it limits the degree to which CBT clinicians can be trained to deliver these treatments, and a particular problem at MGH because referring providers do not have a place to send their patient for CBT services, as trainees constitute a large portion of clinical staff. To address this issue, the current study seeks to document outcomes of CBT interventions delivered by credentialed but not licensed trainees. This information can be used to guide policy and reimbursement guidelines for trainees, as well as promote the ability to disseminate efficacious interventions. Information gained from this project will be used to provide feedback to insurance companies, licensing boards, and mental health community stakeholders regarding decision making re: reimbursement for care provided by supervised trainees. Additionally, this may be used as a pilot study for a comparative effectiveness study comparing trainees to licensed staff psychologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Behavioral Medicine Service are generally individuals with an acute or chronic medical condition or medically related concern with or without an associated DSM-IV psychiatric disorder, as well as adult patients who require assistance with changing health or health-risk behaviors. Patients presenting to the OCD program typically have obsessive compulsive disorder, body dysmorphic disorder, Tourette syndrome, compulsive skin picking, or trichotillomania. Patients presenting to the general CBT program typically have panic disorder, social phobia, generalized anxiety disorder, depression, specific phobia, post traumatic stress disorder, attention deficit hyperactivity disorder, or an eating disorder. Patients at any of the programs have an identifiable behavior or behavioral pattern/ mood problem that they would like to change.
* Age 18 or older
* Ability to provide informed consent and comply with the study procedures
* Ability to complete self-report questionnaires (either written hardcopy or computer-based version) with adequate accommodation, if necessary
* Patients with a PCP at MGH, receiving specialty care at MGH, or employees of MGH.

Exclusion Criteria:

* Exhibit active suicidality (suicidal ideation with intent or plan) to the point that more intensive treatment (i.e. acute hospitalization) is required.
* Active untreated and unstable bipolar disorder (i.e. stable bipolar disorder under care of a psychiatrist is allowed).
* Psychosis.
* Mental retardation.
* Any condition that, after the baseline evaluation, is determined to preclude treatment with cognitive behavioral therapy.
* Received more than 4 sessions of CBT for the target disorder within the past 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The Schwartz Outcome Scale (SOS-10) | at baseline, and at visits 1 through 24, which will occur approximately 1 week apart.
  The Schwartz Outcome Scale (SOS-10) is designed to measure a broad domain of psychological health. It appears to be sensitive to change with treatment. So, we will be measuring whether the total score of this scale changes throughout treatment, i.e., whether the CBT interventions tend to improve psychological health.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Cognitive-Behavioral Therapy and Behavioral Medicine Programs, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Click here to go to the official website of the OCD clinic at Massachusetts General Hospital — http://www.mghocd.org/